CLINICAL TRIAL: NCT02805257
Title: Ahmed Glaucoma Valve Surgery With Mitomycin-C
Acronym: AMCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bascom Palmer Eye Institute (Other); University of North Carolina (Other); University of Colorado, Denver (Other); University of Maryland (Other); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other); Asociación para Evitar la Ceguera en México (Other); Hospital Central Militar (Other Government); Shri Ganesh Vinayak Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#16-18935
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma; Primary Open Angle Glaucoma; Secondary Glaucoma; Neovascular Glaucoma
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Glaucoma, Neovascular | interventions — Mitomycin; Hanks Balanced Salt Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mitomycin-C (Experimental): 0.1 ml of Mitomycin-C 0.4mg/ml injection intraoperatively and twice postoperatively.
  Interventions: Drug: Mitomycin-C; Procedure: Ahmed Glaucoma Valve Implant
- Balanced Salt Solution (BSS) (Placebo Comparator): 0.1ml Balanced Salt Solution injection intraoperatively and twice postoperatively.
  Interventions: Other: Balanced Salt Solution; Procedure: Ahmed Glaucoma Valve Implant

INTERVENTIONS:
Drug: Mitomycin-C — Intraoperative and postoperative injections of mitomycin-c/Mitosol
  Other Names: Mitosol
  Arms: Mitomycin-C
Other: Balanced Salt Solution — Intraoperative and postoperative injections of BSS
  Other Names: BSS
  Arms: Balanced Salt Solution (BSS)
Procedure: Ahmed Glaucoma Valve Implant — Implantation of Ahmed Valve in study eye

SUMMARY:
This study will determine the effectiveness of Mitomycin-C use in the glaucoma surgery Ahmed valve implantation. Approximately 100 patients will be enrolled, with half receiving the Mitomycin-C treatment and the other half receiving placebo treatment.

DETAILED DESCRIPTION:
Glaucoma is a leading cause irreversible blindness worldwide. Glaucoma valve surgeries such as Ahmed valve implantation, which are conventional surgeries performed to control intraocular pressure in eyes, are sometimes associated with complications due to fibrosis. Mitomycin-C is a commonly used antifibrotic agent used in glaucoma surgeries. This study will evaluate the effectiveness of Mitomycin-C injections intraoperatively and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Inadequately controlled glaucoma on maximum tolerated medical therapy with intraocular pressure (IOP) greater than or equal to 18 mm Hg.
* Ahmed Glaucoma Valve (AGV) implantation as the planned surgical procedure.
* For patients in whom 2 eyes are eligible for enrollment, only the first eligible eye to be implanted is enrolled.

Exclusion Criteria:

* Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits.
* Pregnant or nursing women.
* Previous cyclodestruction or glaucoma drainage device (GDD) surgery.
* Patients with nanophthalmos.
* Patients with Sturge-Weber syndrome or other conditions associated with elevated episcleral venous pressure.
* No light perception vision.
* VA <20/200 in non-study eye.
* Need for glaucoma surgery combined with other ocular procedures (i.e. cataract extraction, penetrating keratoplasty, or retinal surgery) or anticipated need for additional ocular surgery.
* Previous scleral buckling procedure or silicone oil present.
* Uveitic glaucoma.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (4):
- University of California, San Francisco, San Francisco, California, United States
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China
- Shri Ganesh Vinayak Eye Hospital, Raipur, Chhattisgarh, India
- Asociación para Evitar la Ceguera en México (APEC), Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
No current plans to share IPD to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Started | 60 | 59
Completed | 53 | 52
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 7 | 6
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS) | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (13.4) | 58.76 (14.8) | 55.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 31 | 34 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Chinese | 9 | 11 | 20
  Ethnicity: Mexican | 51 | 48 | 99
Region of Enrollment [Number; unit: participants]
  China | 9 | 11 | 20
  Mexico | 51 | 48 | 99

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure After Surgery
Description: Goldmann applanation tonometry was used to measure intraocular pressure (IOP) at their one-year after surgery visit, however, for patients with irregular corneal astigmatism, corneal scarring, or corneal edema, which affect accurate measurement, pneumatonometer or Tonopen (Reichert Technologies, Depew, NY) was used. Two consecutive measurements were taken for the study eye. If the 2 measurements differ by 1 mm Hg or less, the IOP for the study eye was the average of the 2 readings. If the 2 measurements differ by 2 mm Hg or more, a third measurement was taken, and the IOP for the study eye was the median of the 3 readings. Efforts were made to schedule follow-up visits at similar time of the day to minimize the effect of diurnal IOP fluctuation. The average IOP and its standard deviation for each arm were calculated based on the individual IOP result obtained using the method described above.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Number analyzed (Participants) | 53 | 52
mmHg | 13.1 (6.3) | 16.2 (6.2)

2. Secondary Outcome: Intraocular Pressure After Surgery
Description: Goldmann applanation tonometry was used to measure intraocular pressure (IOP) at their six-month after surgery visit, however, for patients with irregular corneal astigmatism, corneal scarring, or corneal edema, which affect accurate measurement, pneumatonometer or Tonopen (Reichert Technologies, Depew, NY) was used. Two consecutive measurements were taken for the study eye. If the 2 measurements differ by 2 mm Hg or more, a third measurement was taken, and the IOP for the study eye was the median of the 3 readings. Efforts were made to schedule follow-up visits at similar time of the day to minimize the effect of diurnal IOP fluctuation. The average IOP and its standard deviation for each arm were calculated based on the individual IOP result obtained using the method described above.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Number analyzed (Participants) | 53 | 52
mmHg | 14.6 (8.0) | 16.1 (6.9)

3. Secondary Outcome: Number of Medications Postoperatively
Description: Counted the number of glaucoma drops at six-month after surgery visit. Glaucoma drops are characterized as topical medication used to help lower intraocular pressure.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: glaucoma drops
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Number analyzed (Participants) | 53 | 52
glaucoma drops | 1.2 (0.4) | 1.6 (0.3)

4. Secondary Outcome: Visual Acuity
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity is tested at the six-month after surgery visit. The ETDRS Letter Score is calculated by the number of letters accurately identified at a certain distance, with the range of score being 0-100. An ETDRS letter score of 85 is considered normal vision (equivalent to visual acuity of 20/20), letter scores from 70-84 and 86-100 are considered minimal vision loss and near-normal vision, letter scores from 40-60 are considered moderate visual impairment, and letter scores 0-40 are considered severe visual impairment to total blindness.
Time Frame: 6 months
Population: Unable to report visual acuity data at six months for one Mitomycin-C patient and six Balanced Salt Solution patients due to missing data entry.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Number analyzed (Participants) | 52 | 46
score on a scale | 12.81 (6.98) | 15.33 (6.84)

5. Secondary Outcome: Number of Medications Postoperatively
Description: Counted the number of glaucoma drops at one-year after surgery visit. Glaucoma drops are characterized as topical medication used to help lower intraocular pressure.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: glaucoma drops
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Number analyzed (Participants) | 53 | 52
glaucoma drops | 1.2 (0.3) | 1.6 (0.4)

6. Secondary Outcome: Number of Participants With Intraoperative Complications
Description: Intraoperative complications are characterized as problems that happened during surgery but which were not intended. All complications during surgery were listed and analyzed.
Time Frame: Day of Surgery
Measure: Number; unit: participants
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Number analyzed (Participants) | 53 | 52
participants
  Hyphema | 3 | 5
  Suprachoroidal Hemorrhage | 0 | 0
  Other | 0 | 1

7. Secondary Outcome: Visual Acuity
Description: The Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity is tested at the one-year after surgery visit. The ETDRS Letter Score is calculated by the number of letters accurately identified at a certain distance, with the range of score being 0-100. An ETDRS letter score of 85 is considered normal vision (equivalent to visual acuity of 20/20), letter scores from 70-84 and 86-100 are considered minimal vision loss and near-normal vision, letter scores from 40-60 are considered moderate visual impairment, and letter scores 0-40 are considered severe visual impairment to total blindness.
Time Frame: 1 year
Population: Unable to report visual acuity data at one year for three Mitomycin-C patients and eight Balanced Salt Solution patients due to missing data entry.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Number analyzed (Participants) | 50 | 44
score on a scale | 12.4 (7.33) | 16 (7.78)

8. Secondary Outcome: Number of Participants With Postoperative Complications
Description: Postoperative complications are characterized as problems that happened after surgery but which were not intended. All complications up to the one-year after surgery visit observed were listed and analyzed.
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
Number analyzed (Participants) | 53 | 52
participants
  Tube occlusion | 3 | 1
  Choroidal effusion | 2 | 1
  Suprachoroidal hemorrhage | 1 | 2
  Hyphema | 6 | 7
  Vitreous hemorrhage | 1 | 2
  Shallow Anterior Chamber | 9 | 9
  Corneal edema | 1 | 0
  Endophthalmitis, cystoid macular edema, hypotony maculopathy, tube-K touch, tube erosion, diplopia | 2 | 0
  Other | 8 | 6

ADVERSE EVENTS:
Time Frame: Over 1 Year
Description: In our study protocol, we defined Serious Adverse Events as the following "A SAE is any adverse event that results in any of the following outcomes: death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, or a persistent or significant disability/incapacity."
Arm/Group | Mitomycin-C | Balanced Salt Solution (BSS)
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/52
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52
Other Adverse Events (participants affected / at risk) | 23/53 | 21/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitomycin-C (N=53) | Balanced Salt Solution (BSS) (N=52)
Tube Occlusion (Eye disorders) | 3 | 1
Choroidal Effusion (Eye disorders) | 2 | 1
Suprachoroidal hemorrhage (Eye disorders) | 1 | 2
Hyphema (Eye disorders) | 6 | 7
Vitreous hemorrhage (Eye disorders) | 1 | 2
Shallow Anterior Chamber (Eye disorders) | 9 | 9
Corneal edema (Eye disorders) | 1 | 0
Other (Eye disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT02805257/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT02805257/SAP_001.pdf